CLINICAL TRIAL: NCT00286650
Title: Comparison of Two Different Doses of Paracetamol for Post-Operative Pain Relief
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Otago (Other)
Collaborators: Australian and New Zealand College of Anaesthetists (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Paracetamol
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2006-02-03 (Estimated); Status verified 2004-06

CONDITIONS: Adult Patients Scheduled for 3rd Molar Teeth Extractions
Keywords: Paracetamol

INTERVENTIONS:
Procedure: 3rd molar teeth extraction

SUMMARY:
Paracetamol is commonly used to reduce pain after operations. Recently anaesthetists have been using bigger doses of paracetamol because it has been suggested that bigger doses will work better. However these bigger doses have never been assessed scientifically in adult patients to see if they work better, and it has not been determined at which dose the maximum effect in reducing pain occurs. We We will investigate whether a 90 mg per kg body weight dose works better than a 60 mg per kilogram dose, in reducing pain after wisdom tooth extraction. We will also examine the pharmacokinetics (the way the body removes the drug) of paracetamol, and whether paracetamol changes the way blood clots at these doses. We will also examine whether these doses are safe, by monitoring liver enzymes, and making sure the blood level of paracetamol is not greater than that previously recognised to cause liver disease. The patients will be healthy volunteers scheduled to have wisdom tooth extraction. They will have blood taken at intervals for four hours after having the paracetamol. They will fill in pain scores at the same times they have blood taken.

DETAILED DESCRIPTION:
A randomised, crossover dose-effect trial of paracetamol 60 and 90 mg/kg in third molar surgery

Background Paracetamol is the most widely used analgesic in New Zealand but relatively little is known about its dose effect and concentration effect relationships. It appears that there is greater effect above the currently recommended dose, but the maximal effect has not as yet been described.

Paracetamol is toxic in overdose but the dose at which toxicity becomes apparent is disputed. In the past, the dose at which toxicity may become apparent has been 125 mg/kg/day, but more recently this has been revised upwards to 150 mg/kg/day in children (1). In children it has been proposed that toxicity does not develop following single ingestions of up to 200 mg/kg/day (2).

Paracetamol is metabolised by multiple pathways: urinary excretion of an oral dose is 55% as glucuronide conjugates, 30% as cysteine conjugates, 4% as mercapturic acid and cysteine conjugates (3). The mercapturic and cysteine conjugates are derived from a toxic intermediary metabolite, produced by oxidative metabolism by CYP2E1, and to a lesser degree CYP3A4 and CYP1A2 (4). At doses of up to 1500 mg the metabolism appears to be unchanged but there is no data for doses at or above 90 mg/kg (5). It has been proposed that paracetamol metabolism becomes saturated at higher doses and saturation of sulfation has been observed in rats (6). However saturation of either sulfation or glucuronidation has not been observed in cultured human hepatocytes (6).

In overdose, paracetamol has been observed to inhibit the activity of vitamin-K dependent clotting factors, in particular functional factor VII (7). This may explain the interaction between paracetamol and warfarin.

Aims

* To describe the dose and effect relationship for paracetamol
* To describe the concentration and effect relationship for paracetamol
* To examine the changes in metabolism of paracetamol with escalating doses
* To examine the effect of paracetamol on functional factor VII (effect on coagulation mechanism) with increasing dose

Methods

Subjects:

Eighteen healthy adults, male or female, aged 18 to 50 years scheduled for removal of bilateral, impacted, lower wisdom teeth will be recruited for the trial in the dental school.

Exclusion criteria:

* Intolerance to oral medication
* Taking paracetamol and unable to abstain prior to the study
* Hypersensitivity to paracetamol
* Liver or renal failure
* Pregnancy
* Breast feeding
* Poor nutritional status, eating disorder, or Body Mass Index (BMI) less than 16
* Weight greater than 87 kg
* Anticonvulsant medication
* Chronic ethanol abuse
* H/o bleeding disorders

Participants will be instructed to avoid all non-essential medications, paracetamol, alcohol, herbal medicines and recreational drugs for 72 hours prior to the study and are required to fast for three hours prior to the study.

Demographic data Demographic data including height, weight and age will be recorded for each patient. Medications pre-, peri- and post-operatively will be recorded. Regular use of alcohol, caffeinated beverages and smoking will be recorded.

Treatment:

The patients will be fasted for three hours prior to the procedure. An intravenous line will be inserted and intravenous midazolam administered, with the dose titrated to sedative effect; use of sedation, oral or intravenous, for third molar extractions is a common practice in dentistry. Local anaesthetic (2% Lignocaine with adrenaline 1/80000) will be administered at the commencement of the procedure. The paracetamol will be administered as capsules, made by the Pharmacy Dept of the University of Otago 30 minutes prior to the procedure. Dosing will be observed.

Rndomised, double blind, cross over design will be used for each side for the surgery. Both the side of extraction and the treatment will be randomised.

During the procedure the patients will be observed by using pulse oximetry and blood pressure. The patients will be requested to stay at the dental school for 4 hours after the paracetamol dosing.

If the patient should require additional pain relief, they will be given codeine 30 mg or diclofenac 50 mg. The patients will be instructed to avoid additional doses of paracetamol for 48 hours. Further analgesia on subsequent days will be provided with NSAIDs (diclofenac) and/ or codeine phosphate In appropriate doses Prophylactic antibiotics will be used where necessary according to usual treatment practice.-

Samples:

Blood will be collected at times: 0, 15, 30, 60, 90, 120, 180, 240, 480 minutes through the cannula already in place in the standard manner. (Note time 0 is the time of paracetamol dosing). 3-6 mL of blood is collected on each occasion and then transferred into a 6 mL heparinised saline vacutainer®. These will be spun in an Eppendorf® Centrifuge 5810R at 4000 g for 5 minutes. Plasma will be removed and transferred into a 2 mL microtube (Eppendorf® safe lock) prior to freezing at -20°C. The catheter line and extension will be kept patent using heparinised saline (10 IU/ mL) flushes.

Urine collected from: (pass urine at time 0 and discard), 0 to 120, 120 to 240 and 240 to 480 minutes. Urine volume will be measured and recorded. An aliquot of urine from each time interval will be stored at -200C prior to assay.

Blood will also be collected at 0 and 24 hours for ALT, AST, PT and clotting factors.

An additional sample of blood will be collected at four hours after administration of paracetamol forserum paracetamol level estimation. . If this level is greater than the treatment threshold on the New Zealand Poisons Centre Substance Database, the patient will be treated with n-acetylcysteine by the standard treatment protocol as soon as possible.

Pain score:

Visual analogue pain score (0-100 mm scale) will be recorded at 0, 30, 60, 90, 120, 150, 180, 210, 240, 480 minutes and at 24 hours after the end of surgery. Mouth opening (trismus) will be assessed at 0 and 24 hours.

Analytical methods:

Urine:

All samples were analysed using high performance liquid chromatography (HPLC) to determine the concentrations of paracetamol and its metabolites, paracetamol glucuronide, paracetamol cysteine, paracetamol sulphate and paracetamol mercapturate. Urine samples were prepared for HPLC by centrifuging at 2000rpm and then diluting the supernatent 1 in 10 with mobile phase. This was injected directly onto an Aqua C18 reversed phase column, 250mm x 4.6mm i.d. with a 5 micron pore size (Phenomenex) via a C18, 5 micron guard column. The mobile phase used was 7% acetonitrile - 93% orthophosphoric acid (20mM pH 6.7) at a flow rate of 1ml/min using a Shimadzu LC10-AT pump and a Shimadzu SPD-10AV ultraviolet absorbance detector operating at 254nm. Calibration curves were constructed for each of the metabolites and paracetamol in blank urine using the peak area and were linear over the range 0.05 - 5mM. The method was found to be reproducible with a coefficient of variation of 2.6%. The metabolites of paracetamol; glucuronide, cysteine, sulphate, mercapturate and paracetamol itself eluted in 3.9, 8, 10.2, 12.2 and 13.4 minutes respectively. Reference samples of paracetamol cysteine, sulphate and mercapturate were kindly supplied by Dr Anthony R. Temple MD, McNeil Consumer Healthcare, Camp Hill Road, Fort Washington, Pennsylvania, USA.

Sample size calculation:

Previous studies of dental pain have indicated a maximum intensity of pain at around 8 hours following third molar extractions. On a 100 mm visual analogue scale the mean (S.D.) pain score was 40.9 (24.4). At a pain score of 27.3 the S.D. was 17.2. We estimate that 17 patients are required for a power of 80% and a 50% decrease in pain.

Ethical issues The fee for surgery will be waived for the participants. There will be no other financial inducement. Paracetamol is known to cause hepatotoxicity and fatality in overdosage. These effects have not been reported with single ingestions of less than 150 mg/kg.

The patient will be undergoing a dental procedure and there will be the normal risks associated with such procedures.

1. National Poisons Centre New Zealand. toxinz. In; 2001.
2. Mohler C, Nordt SP, Williams SR, Manoguerra AS, Clark RF. Prospective evaluation of mild to moderate pediatric acetaminophen exposures. Ann Emerg Med 2000;37(1):114-116.
3. Prescott LF. Kinetics and metabolism of paracetamol and phenacetin. Br J Clin Pharmacol 1980;10(Suppl 2):291S-298S.
4. Dai Y, Cederbaum AI. Cytotoxicity of acetaminophen in human cytochrome P4502E1-transfected HepG2 cells. J Pharmacol Exp Ther 1995;273(3):1497-1505.
5. Steventon GB, Mitchell SC, Waring RH. Human metabolism of paracetamol (acetaminophen) at different dose levels. Drug Metabol Drug Interact 1996;13(2):111-117.
6. Kane RE, Li AP, Kaminski DR. Sulfation and glucuronidation of acetaminophen by human hepatocytes cultured on Matrigel and type 1 collagen reproduces conjugation in vivo. Drug Metab Dispos 1995;23(3):303-307.
7. Whyte IM, Buckley NA, Reith DM, Goodhew I, Seldon M, Dawson AH. Acetaminophen causes an increased International Normalized Ratio by reducing functional factor VII. Ther Drug Monit 2000;22(6):742-748.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen healthy adults, male or female, aged 18 to 50 years scheduled for removal of bilateral, impacted, lower wisdom teeth will be recruited for the trial in the dental school.

Exclusion Criteria:

* Intolerance to oral medication
* Taking paracetamol and unable to abstain prior to the study
* Hypersensitivity to paracetamol
* Liver or renal failure
* Pregnancy
* Breast feeding
* Poor nutritional status, eating disorder, or Body Mass Index (BMI) less than 16
* Weight greater than 87 kg
* Anticonvulsant medication
* Chronic ethanol abuse
* H/o bleeding disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2005-05; Study Completion 2005-10

PRIMARY OUTCOMES:
Any difference in effectiveness between the 2 dosage schedules

SECONDARY OUTCOMES:
Any difference in safety between the 2 dosage schedules

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Zacharias, Dr, Principal Investigator — Dunedin School of Medicine, Dunedin, New Zealand
Locations (1):
- School of Dentistry, University of Otago, Dunedin, Otago, New Zealand